CLINICAL TRIAL: NCT00712556
Title: Positron Emission Tomography Study in Patients With Non-Hodgkin Lymphoma
Brief Title: PET Study in Patients With Non-Hodgkin Lymphoma
Status: Completed | Type: Observational
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Responsible Party: Principal Investigator, Adetola A. Kassim, Associate Professor of Medicine; Clinical Director, Sickle Cell Anemia Program; Hematologist/Oncologist, Vanderbilt-Ingram Cancer Center
Other Study IDs: VICC BMT 0828; VU-VICC-BMT-0828; VU-VICC-080426
Record Dates: First submitted 2008-07-09; First posted 2008-07-10 (Estimated); Last update posted 2013-02-26 (Estimated); Status verified 2013-02

CONDITIONS: Lymphoma
Keywords: stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III small lymphocytic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent childhood large cell lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; recurrent mycosis fungoides/Sezary syndrome; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; NC stage II adult immunoblastic large cell lymphoma; NC stage II adult lymphoblastic lymphoma; NC stage II grade 1 follicular lymphoma; NC stage II grade 2 follicular lymphoma; NC stage II grade 3 follicular lymphoma; NC stage II mantle cell lymphoma; NC stage II marginal zone lymphoma; NC stage II small lymphocytic lymphoma
MeSH Terms: conditions — Lymphoma; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Flourine 18-fluorodeoxyglucose PET: PET using fluorine 18-fluorodeoxyglucose to image cancer tumors
  Interventions: Radiation: fluorine 18-fludeoxyglucose positron emission tomography

INTERVENTIONS:
Radiation: fluorine 18-fludeoxyglucose positron emission tomography — fluorine 18-fludeoxyglucose is a radioactive isotope used in PET to detect cancer tumors
  Other Names: fluorine 18-fludeoxyglucose PET

SUMMARY:
RATIONALE: Diagnostic procedures, such as fluorine 18-fludeoxyglucose positron emission tomography (PET) scans, may help doctors predict a patient's response to treatment and help plan the best treatment.

PURPOSE: This phase I trial is studying fluorine 18-fludeoxyglucose PET scan to see how well it predicts outcomes in patients who have undergone high-dose chemotherapy and autologous stem cell transplant for non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine if a fluorine 18-fludeoxyglucose positron emission tomography scan, performed as early as day 30 after high-dose chemotherapy and autologous stem cell transplantation, may be useful in identifying patients with non-Hodgkin lymphoma who may benefit from early interventions, including reduced intensity stem cell transplantation or additional therapy, to preempt disease relapse and improve overall survival.

OUTLINE: Conventional imaging, biopsy, and clinical examination findings are reviewed to determine patient clinical outcome (e.g., complete remission, disease progression/relapse, or death related to the primary disease).

ELIGIBILITY:
Inclusion Criteria:

DISEASE CHARACTERISTICS:

* Diagnosis of non-Hodgkin lymphoma
* Has undergone high-dose chemotherapy followed by autologous stem cell transplantation at Vanderbilt University between March 1997 and August 2005

  * Has undergone fluorine 18-fludeoxyglucose PET within 70 days prior to and/or at approximately 30 days and 100 days after high-dose chemotherapy and autologous stem cell transplantation

Exclusion Criteria:

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with non-Hodgkin lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2008-05; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Correlation of sensitivity, specificity, positive predictive value, and negative predictive value of fluorine 18-fludeoxyglucose positron emission tomography scan with with patients' clinical outcomes. | from the date of stem cell transplant to date of clinical disease progression or to date of last follow-up

SECONDARY OUTCOMES:
Progression-free survival | from date of stem cell transplant to date of clinical disease progression or date of last follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Adetola A. Kassim, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (3):
- United States (3):
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Franklin, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee